CLINICAL TRIAL: NCT02548000
Title: Muscle and Vascular Adaptations Induced by Resistance Training in Elderly Diabetic Type 2
Brief Title: Diabetes Resistance Training Adaptations in Elderly
Acronym: DRTAE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 150257
Record Dates: First submitted 2015-08-25; First posted 2015-09-14 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resistance training (Experimental): Resistance training will be performed three times a week, for 12 weeks, composed by 12 resistance exercises for all body muscles with 2-3 series and 12-8 repetitions in each exercise.
  Interventions: Other: Resistance training
- Stretching control (Active Comparator): The control group will perform one stretching session a week.
  Interventions: Other: Stretching control

INTERVENTIONS:
Other: Resistance training — The resistance training will be compound by 12 exercises for all body muscles, performed three times per week. The intensity of training will be measure by maximum repetitions from 12 until 8 repetitions with 2-3 series. The loads will increase for keep the maximum strength as the capacity of patients. The blood pressure and the casual glycemic will be measure before and after the training in each session. Before to start the exercises, patients will perform a warming on treadmill for 10 minutes and after the training will perform some stretching exercises for muscles groups trained.
  Arms: Resistance training
Other: Stretching control — The stretching session will be composed by stretching and joint mobilization exercises for all body muscles and will happen only one time per week.
  Arms: Stretching control

SUMMARY:
This study aims to verify the effects of resistance training on neuromuscular, vascular and functional adaptations of elderly diabetics type 2. Half of participants will be the intervention group that will perform resistance training, while the other half will be the control group that will perform stretching sessions.

DETAILED DESCRIPTION:
Resistance training may be an interesting strategy to fight diabetes deleterious conditions, as it is known to increase muscle mass and quality, strength, functional capacity, vascular health, and decrease inflammation status and blood lipids, besides leading to improves in glycemic control. To test this hypothesis, 42 diabetic patients will be recruited and randomized to two groups that will be evaluated before and after 12 weeks of both intervention or control period. The resistance training group will perform all body resistance exercises three times per week, while the control group will perform a stretching session one time per week.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* 60 yers and older
* HbA1c > 6,5%
* BMI from 18,5 kg/m2 - 34,9 kg/m2

Exclusion Criteria:

* Current smoking
* Insulin users
* Hypertension uncontrolled
* Diabetic neuropathy
* Diabetic retinopathy
* Diabetic nephropathy
* Peripheral amputations
* Clinical depression
* Myocardial infarction (within past 6 months)
* Any unstable chronic condition
* Muscle-skeletal complications that limit the practice of the exercises

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Quadriceps Muscle Quality measure by echo intensity | 12 weeks
  Echo intensity is a grey scale for analyse the image that ranging from 0 (black) to 255 (white).

SECONDARY OUTCOMES:
Functional capacity measure by stair climb test. | 12 weeks
  Total time, as fast as possible, to climb 10 steps.
Quadriceps muscle strength measured by one repetition maximum (1RM) test. | 12 weeks
  1RM is a maximum load lifted, reported in kg, during the knee extension.
Visceral adipose tissue measured by ultrasonography | 12 weks
  Visceral adipose tissue (VAT) thickness measured by ultrasonography. The VAT thickness is considered from the back of the subcutaneous tissue until the anterior part of the aorta. It is reported in mm.
Muscle thickness measured by ultrasonography | 12 weeks
  Muscle thickness measured by ultrasonography takes into account the superior fascia of the muscle and the distance until the inferior fascia. It is reported in mm.
Inflammation status estimated by tumor necrosis factor alpha (TNF-α ) and C reactive protein (CRP) | 12 weeks
  TNF-α will be evaluated by specific commercial kit and CRP will be measured in a regular laboratorial equipment (COBAS C111).
Lipid profile | 12 weeks
  HDL, LDL, total cholesterol and triglycerides will be measured in a regular laboratorial equipment (COBAS C111)
Glycemic profile | 12 weeks
  Blood glycated hemoglobin and glucose will be measured in a regular laboratorial equipment (COBAS C111)
Endothelial function measured by ultrasonography | 12 weeks
  Endothelial function estimated by the response of endothelial cells for hyperemia.
Quadriceps Muscle Quality measure by specific tension | 12 weeks
  Specific tension is the ratio between muscle strength and muscle mass.
Functional capacity measure by time up and go test | 12 weeks
  Time to get up from the chair walk around the marker (3 m) and return to the sitting position, as fast as possible.
Functional capacity measure by sit-to-stand-up test | 12 weeks
  The time, as fast as possible, to stand and sit on the chair 10 times.
Quadriceps muscle power capacity measure by rate of torque development. | 12 weeks
  The rate torque development is a slope of torque/time curve.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre S Dias, phd, Study Director — Hospital de Clinicas de Porto Alegre
Locations (2):
- Brazil (2):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Federal University of Rio Grande do Sul, Physical Education School, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: Undecided